CLINICAL TRIAL: NCT03694886
Title: The Effect of Tablet Size on Cognitive Performance: A Randomized Control Trial Using Caffeine
Brief Title: The Effect of Tablet Size on Cognitive Performance Caffeine
Acronym: CaC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 18-1086
Record Dates: First submitted 2018-10-01; First posted 2018-10-03 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Placebo Effect
MeSH Terms: interventions — Sugars

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of four groups:
  1) 90 mg caffeine with a 1 mm diameter sucrose pillule; 2) no caffeine with the small sucrose pillule; 3) 90 mg caffeine with a 5 mm sucrose pillule; 4) no caffeine with the large sucrose pillule.
Who Masked: Participant
Masking Description: Participants will not be made aware if they have or have not received caffeine to not bias results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Caffeine with small sucrose pill (Active Comparator): Participants will be given one dose of 90 milligrams caffeine anhydrous dissolved in 8 ounces of water and a 1 mm sucrose pill to consume in 10 minutes. After 30 minutes post-administration, the cognitive tests will be administered.
  Interventions: Drug: Caffeine Anhydrous with small sucrose pill
- Caffeine with large sucrose pill (Active Comparator): Participants will be given one dose of 90 milligrams caffeine anhydrous dissolved in 8 ounces of water and a 5 mm sucrose pill to consume in 10 minutes. After 30 minutes post-administration, the cognitive tests will be administered.
  Interventions: Drug: Caffeine Anhydrous with large sucrose pill
- No caffeine with small sucrose pill (Placebo Comparator): Participants will be given 8 ounces of water and a 1 mm sucrose pill to consume in 10 minutes. After 30 minutes post-administration, the cognitive tests will be administered.
  Interventions: Other: Placebo - small sucrose pill
- No caffeine with large sucrose pill (Placebo Comparator): Participants will be given 8 ounces of water and a 1 mm sucrose pill to consume in 10 minutes. After 30 minutes post-administration, the cognitive tests will be administered.
  Interventions: Other: Placebo - large sucrose pill

INTERVENTIONS:
Drug: Caffeine Anhydrous with small sucrose pill — caffeine anhydrous that has been weighed out to 90 mg per dose presented with a 1 mm sucrose pillule
  Other Names: pure caffeine powder
  Arms: Caffeine with small sucrose pill
Other: Placebo - large sucrose pill — sucrose pillules of 5 mm diameter will be given to all participants in the large pill groups
  Other Names: sugar pill
  Arms: No caffeine with large sucrose pill
Drug: Caffeine Anhydrous with large sucrose pill — caffeine anhydrous that has been weighed out to 90 mg per dose presented with a 5 mm sucrose pillule
  Other Names: pure caffeine powder
  Arms: Caffeine with large sucrose pill
Other: Placebo - small sucrose pill — sucrose pillules of 1 mm diameter will be given to all participants in the small pill groups
  Other Names: sugar pill
  Arms: No caffeine with small sucrose pill

SUMMARY:
This study aims to assess if tablet size, due to placebo effect, alters participants' performance on cognitive tests after consuming caffeine. Participants will be randomly assigned to one of four groups: 1) 90 mg caffeine with a 1 mm diameter sucrose pillule; 2) no caffeine with the small sucrose pillule; 3) 90 mg caffeine with a 5 mm sucrose pillule; 4) no caffeine with the large sucrose pillule.

DETAILED DESCRIPTION:
Background: A capsule's physical design (e.g. shape, size, and color) affects individuals' perception of drug efficacy; that is, how well a drug is likely to work. The goal of this study is to assess the effects tablet size may have on participant's performance on cognitive testing since research has found differences between preparation methods. Method: 120 participants will be randomly assigned to one of four groups: 1) 90 mg caffeine with a 1 mm diameter sucrose pillule; 2) no caffeine with the small sucrose pillule; 3) 90 mg caffeine with a 5 mm sucrose pillule; 4) no caffeine with the large sucrose pillule. Participants will consume the designated placebo tablet with water (caffeinated or non-caffeinated); then, participants will provide weekly caffeine intake and complete the neutral portion of Velten's Mood Induction Procedure until 30 minutes have passed to allow for caffeine activation. Participants will complete the Stroop test, Trial Making Tests A and B, and the Rey Auditory Verbal Learning Test. Previous literature, as far as the author knows, relied on evaluating drug efficacy based on appearance alone. This study aims to assess if tablet size, due to placebo effect, alters participants' performance on cognitive tests after consuming caffeine.

ELIGIBILITY:
Inclusion Criteria:

* Fluent in written and spoken English
* Ability to see color
* No uncontrolled high blood pressure
* No allergies to caffeine or sucrose
* No history of heart disease
* No untreated anxiety or depression
* Non-pregnant
* No caffeine consumed the day of participation

Exclusion Criteria:

* Not fluent in written and/or spoken English
* Uncontrolled high blood pressure
* Color-blindness
* Allergies to caffeine and/or sucrose
* History of heart disease
* Untreated anxiety or depression
* Pregnant
* Consumed caffeine on the day of participation

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2018-10-31 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Stroop Color test | Within 90 minutes of receiving informed consent. Actual task time: approximately 1.5 minutes
  Measures processing speed. 100-item, time-trial task where participants read the color of printed items on the task paper as quickly as possible for 45 seconds. Scores are measured in the number of correct responses within the allotted time.
Stroop Word test | Within 90 minutes of receiving informed consent. Actual task time: approximately 1.5 minutes
  Measures processing speed. 100-item, time-trial task where participants read color names printed on the task paper as quickly as possible for 45 seconds. Scores are measured in the number of correct responses within the allotted time.
Trail Making task A | Within 90 minutes of receiving informed consent. Actual task time: approximately 2 minutes
  Measures processing speed. 25 item, time-trial task where participants must connect numbers in order as quickly as possible. Scores are measured by the amount of time (in seconds) for participants to complete the task.

SECONDARY OUTCOMES:
Stroop Color-and-Word test | Within 90 minutes of receiving informed consent. Actual task time: approximately 2 minutes
  Measures processing speed. 100-item, time-trial task where participants must read the color of the ink instead of color names printed on the task paper as quickly as possible for 45 seconds. Scores are measured in the number of correct responses within the allotted time.
Trail Making task B | Within 90 minutes of receiving informed consent. Actual task time: approximately 3 minutes
  Measures processing speed. 25 item, time-trial task where participants must connect numbers and letters in order (e.g. 1-A-2-B, etc.) as quickly as possible. Scores are measured by the amount of time (in seconds) for participants to complete the task.
Rey Auditory Verbal Learning test | Within 90 minutes of receiving informed consent. Actual task time: approximately 40 minutes
  Measures memory. 30-item, 2 section task where participants are read 15 words and asked to recall as many words as possible in the first section. A second set of 15 words is then introduced and participants recall those. The second section consists of revisiting the original set of words and recalling as many of those. Scores are measured by the total words remembered in section one, and another score for the total intrusions from the second list into the recall of section two.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Hernandez Altamirano, Principal Investigator — Undergraduate honors student
Locations (1):
- University of Colorado Denver, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beaumont R, Cordery P, Funnell M, Mears S, James L, Watson P. Chronic ingestion of a low dose of caffeine induces tolerance to the performance benefits of caffeine. J Sports Sci. 2017 Oct;35(19):1920-1927. doi: 10.1080/02640414.2016.1241421. Epub 2016 Oct 20. PMID 27762662
- [Background] Buckalew LW, Coffield KE. An investigation of drug expectancy as a function of capsule color and size and preparation form. J Clin Psychopharmacol. 1982 Aug;2(4):245-8. PMID 7119132
- [Background] Champlin SE, Pasch KE, Perry CL. Is the Consumption of Energy Drinks Associated With Academic Achievement Among College Students? J Prim Prev. 2016 Aug;37(4):345-59. doi: 10.1007/s10935-016-0437-4. PMID 27236788
- [Background] Cole JS. A survey of college-bound high school graduates regarding circadian preference, caffeine use, and academic performance. Sleep Breath. 2015 Mar;19(1):123-7. doi: 10.1007/s11325-014-0976-y. Epub 2014 May 1. PMID 24788599
- [Background] Czerniak E, Davidson M. Placebo, a historical perspective. Eur Neuropsychopharmacol. 2012 Nov;22(11):770-4. doi: 10.1016/j.euroneuro.2012.04.003. Epub 2012 May 18. PMID 22608298
- [Background] Franzen MD, Tishelman AC, Sharp BH, Friedman AG. An investigation of the test-retest reliability of the Stroop Color-Word Test across two intervals. Arch Clin Neuropsychol. 1987;2(3):265-72. PMID 14589618
- [Background] Geuter S, Koban L, Wager TD. The Cognitive Neuroscience of Placebo Effects: Concepts, Predictions, and Physiology. Annu Rev Neurosci. 2017 Jul 25;40:167-188. doi: 10.1146/annurev-neuro-072116-031132. Epub 2017 Apr 7. PMID 28399689
- [Background] Hammond DC. A review of the history of hypnosis through the late 19th century. Am J Clin Hypn. 2013 Oct;56(2):174-91. doi: 10.1080/00029157.2013.826172. PMID 24665818
- [Background] Ibrahim IR, Ibrahim MI, Al-Haddad MS. The influence of consumers' preferences and perceptions of oral solid dosage forms on their treatment. Int J Clin Pharm. 2012 Oct;34(5):728-32. doi: 10.1007/s11096-012-9667-6. Epub 2012 Jun 29. PMID 22744843
- [Background] Kinirons MT, O'Mahony MS. Drug metabolism and ageing. Br J Clin Pharmacol. 2004 May;57(5):540-4. doi: 10.1111/j.1365-2125.2004.02096.x. PMID 15089805
- [Background] Lessard, M. D. (1993). Study of the Velten Mood Induction Procedure and the measurement of mood. Graduate Student Theses, Dissertations, & Professional Papers. 4973. https://scholarworks.umt.edu/etd/4973
- [Background] Magalhaes, S. d. S., Malloy-Diniz, L. F., & Hamdan, A. C. (2012). Validity convergent and reliability test-retest of the rey auditory verbal learning test. Clinical Neuropsychiatry: Journal of Treatments Evaluation, 9(3), 129.
- [Background] Nehlig A, Daval JL, Debry G. Caffeine and the central nervous system: mechanisms of action, biochemical, metabolic and psychostimulant effects. Brain Res Brain Res Rev. 1992 May-Aug;17(2):139-70. doi: 10.1016/0165-0173(92)90012-b. PMID 1356551
- [Background] Overgaard AB, Hojsted J, Hansen R, Moller-Sonnergaard J, Christrup LL. Patients' evaluation of shape, size and colour of solid dosage forms. Pharm World Sci. 2001 Oct;23(5):185-8. doi: 10.1023/a:1012050931018. PMID 11721676
- [Background] Pasman WJ, Boessen R, Donner Y, Clabbers N, Boorsma A. Effect of Caffeine on Attention and Alertness Measured in a Home-Setting, Using Web-Based Cognition Tests. JMIR Res Protoc. 2017 Sep 7;6(9):e169. doi: 10.2196/resprot.6727. PMID 28882811
- [Background] Pettit ML, DeBarr KA. Perceived stress, energy drink consumption, and academic performance among college students. J Am Coll Health. 2011;59(5):335-41. doi: 10.1080/07448481.2010.510163. PMID 21500050
- [Background] Ross, S., & Buckalew, L. W. (1979). On the agentry of placebos. American Psychologist, 34(3), 277-278. 10.1037/0003-066X.34.3.277
- [Background] Scientific Opinion on the substantiation of health claims related to caffeine and increased fat oxidation leading to a reduction in body fat mass (ID 735, 1484), increased energy expenditure leading to a reduction in body weight (ID 1487), increased alert. (2011). EFSA Journal, 9(4), 2054. doi:10.2903/j.efsa.2011.2054
- [Background] Smith SR, Servesco AM, Edwards JW, Rahban R, Barazani S, Nowinski LA, Little JA, Blazer AL, Green JG. Exploring the validity of the comprehensive trail making test. Clin Neuropsychol. 2008 May;22(3):507-18. doi: 10.1080/13854040701399269. Epub 2007 Jun 18. PMID 17853128

DOCUMENTS (2):
  • Informed Consent Form (2018-09-20): https://cdn.clinicaltrials.gov/large-docs/86/NCT03694886/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2018-07-09): https://cdn.clinicaltrials.gov/large-docs/86/NCT03694886/Prot_SAP_001.pdf